CLINICAL TRIAL: NCT07265622
Title: A Phase I/II Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of 7MW4911 in Patients With Advanced Solid Tumors
Brief Title: First-in-human Study of 7MW4911 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7MW4911-CP102
Record Dates: First submitted 2025-11-16; First posted 2025-12-05 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 7MW4911 (Experimental)
  Interventions: Drug: 7MW4911

INTERVENTIONS:
Drug: 7MW4911 — 7MW4911 for IV infusion of various dose strengths administered

SUMMARY:
This is the first-in-human study of 7MW4911 in Chinese patients, to investigate its prelimary safety and efficacy in patients with Advanced Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18~75.
2. ECOG 0-1.
3. Life expectancy ≥ 3 months.
4. Participants with pathologically (histologically or cytologically) confirmed advanced solid tumors.
5. Disease progression after the most recent treatment regimen.
6. At least one measurable lesion according to RECIST v1.1.
7. Provision of archival tumor tissue or fresh biopsy.
8. Adequte hematologic funciton, liver function and renal function.
9. Comply with contraceptive requirements.

Exclusion Criteria:

1. Other concurrent malignancy in the recent 3 years except for adequately treated carcinoma in situ.
2. Active, untreated or symptomatic CNS metastasis.
3. Effusions that require frequent drainage.
4. Patients with active autoimmune disease, except for type I diabetes, hypothyroidism and other autoimmune disease that does not require systemic treatment.
5. Severe respiratory disease that required hospitalization in the last 28 days.
6. Significant and uncontrolled cardiovascular disease or events in the 6 months prior to study drug administration.
7. Poorly controlled blood glucose with fasting blood glucose above 10 mmol/L.
8. Recipient of allogeneic stem cell transplant or organ transplant
9. Active HIV or hepatitis B/C infection. Infection requiring systemic IV in the 14 days prior to study drug administration.
10. Experiencing toxicities from prior anti-cancer therapies that have not recovered to CTCAE grade 0-1, except for alopecia and endocrinopathies.
11. Prohibited treatment and treatment that requires washout period: (1) Has received another Topo-I payload ADC, and/or another CDH17 targeting therapy. (2) Received other cancer therapy within 5 half-lives or 21 days prior to study drug administration. (3) Major surgeries within 28 days prior to study drug administration. (4) Investigational therapy within 28 days prior to study drug administration. (5) Systemic treatment with immunosuppressive agents within 28 days prior to first drug administration. Physiological dose of glucocorticoid, topical glucocorticoid are allowed. (6) Use of strong CYP3A4 inhibitor or inducer.
12. Known hypersensitivity to 7MW4911 or components of the formulation.
13. Abuse of narcotic or psychoactive drugs.
14. Pregnant or breastfeeding women.
15. Other circumstances or conditions where the investigator judges to be unsuitable for study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-12 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and rates of adverse events | Up to approximately 2 years
  To assess the safety and tolerability of 7MW4911 in patients with advanced colorectal cancer and other advanced gastrointestinal tumors
Maximum tolerated dose (MTD), recommended expansion dose (RED) and the recommended phase II dose (RP2D) | Up to approximately 2 years
  To determine the maximum tolerated dose (MTD) and recommended expansion dose (RED) or the recommended phase II dose (RP2D)

SECONDARY OUTCOMES:
Objective response rate | Up to approximately 2 years
  Proportion of patients whose turmor response meet the criteria of complete response or partial response
Progression-free survival | Up to approximately 2 years
  Duration in months from treatment to disease progression or death from any cause, whichever occurs first.
Immunogenicity | Up to approximately 2 years
  Incidence and rates of ADA
Tmax | Up to 3 months
  Time to maximum concentration of 7MW4911 in blood
Cmax | Up to 3 months
  Maximum concentration of 7MW4911 in bloood
t1/2 | Up to 3 months
  Time to decrease of 7MW4911 concentration by 50% in blood
Area under the curve | Up to 3 months
  Area Under the Plasma Concentration-Time Curve from Time Zero to Last Measurable Concentration (AUC0-t)

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China